CLINICAL TRIAL: NCT06644846
Title: A Prospective Study of Spatially Fractionated Radiation Treatment Using Rapid Rod Technique for Gynaecological Cancers
Brief Title: Spatially Fractionated Radiation Treatment for Gynaecological Cancers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Dr Supriya Sastri, Tata Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC IEC III 900965
Record Dates: First submitted 2024-07-12; First posted 2024-10-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cervical Cancer; Gynecologic Cancer; Recurrent Cancer
Keywords: Cervical cancer; Cancer; Recurrence; Spatially fractionated radiotherapy; Rapid rod
MeSH Terms: conditions — Uterine Cervical Neoplasms; Recurrence; Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention type: Spatially Fractionated Radiation Therapy (SFRT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SFRT arm (Experimental): This is a single arm phase II study. All patients will receive the planned intervention ie. spatially fractionated radiation therapy using rapid rod technique.
  Interventions: Radiation: Spatially fractionated radiation therapy

INTERVENTIONS:
Radiation: Spatially fractionated radiation therapy — Spatially fractionated" radiation therapy (SFRT) enables delivery of high-dose radiation to discrete sub-volumes inside a tumour target while restricting the remainder of the target to a safer lower dose. This technique results in generation of intentionally heterogeneous dose distribution with spatial areas of "hot" and "cold" spots within the tumour, thereby sparing nearby organs at risk.

SUMMARY:
This is a prospective study to evaluate in-field disease control, survival and late toxicity in patients with cervical cancer or pelvic recurrence treated with spatially fractionated RT.

The study will include patients with primary cervical cancer or pelvic recurrence not suitable for brachytherapy in view of anticipated or actual suboptimal target coverage due to aberrant anatomy or large residual disease at the time of brachytherapy.

DETAILED DESCRIPTION:
Patients will be treated with spatially fractionated radiation therapy (SFRT) after EBRT completion to a dose of 25-30 Gy in 5-6 fractions in the primary setting. For patients receiving re-irradiation, 20-25 Gy in 4-5 fractions will be delivered with SFRT, which however may be individualised to match with clinical practice in the re-RT setting. Total EQD2 Gy for organs at risk will be matched to brachytherapy.

The study will be conducted at Tata Memorial Hospital, Mumbai and Advanced Centre for Treatment, Research and Education In Cancer (ACTREC), Navi Mumbai.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cervical cancer post EBRT, with expected suboptimal brachytherapy dose coverage due to-

   1. Aberrant uterine or pelvic anatomy leading to difficulty in localization of the cervical OS or negotiation of the uterine canal accurately by two independent clinicians in up to two procedures.
   2. Large residual disease at the time of brachytherapy with anticipated suboptimal target coverage either determined in clinic based on pre-brachytherapy imaging or at dose planning (e.g. figure 2).
   3. Very narrow vaginal canal not accommodating even the smallest intracavitary or vaginal cylinder applicators.
2. Patients with inoperable endometrial cancer not suitable for anaesthesia or have anticipated suboptimal coverage of target volume at brachytherapy as identified on pre-brachytherapy imaging obtained after EBRT.
3. Patients with large pelvic recurrences after surgery and/or (chemo) radiation, not amenable to surgical salvage or brachytherapy after salvage EBRT due to reasons specified in item 1.
4. Patients with contraindications to anaesthesia for brachytherapy with sufficient risk of on-table or post procedure adverse events.

Exclusion Criteria:

1. Any pre-existing fistula in bladder or rectum.
2. Pelvic prosthesis.
3. Refusal to provide consent.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
In-field control | 1-year
  To evaluate in-field local control patients with cervical cancer or pelvic recurrence treated with spatially fractionated RT

SECONDARY OUTCOMES:
Progression-free and overall survival | 2-years
  To evaluate progression free and overall survival from the date of end of treatment upto 2 years
Late grade 2 or higher genitourinary and gastrointestinal toxicities. | > 90 days
  To evaluate grade 2 or higher genitourinary and gastrointestinal toxicities from the date of end of treatment upto 90 days
To compare SFRT in-silico dose volume parameters with proton beam plans | 1-year
  To compare dose volume parameters of SFRT plans with proton beam plans, created on the same datasets.
To obtain biopsy tissue for translational research before and after SFRT | 1-year
  Programmed cell death ligand 1 (PD-L-1) expression will be studied
To study overall response in reference to PET FDG and Hypoxia imaging at baseline and before SFRT | 1-year
  To evaluate overall response based on PET-FDG and hypoxia markers at baseline and before SFRT

CONTACTS AND LOCATIONS:
Locations (1):
- ACTREC Tata Memorial Centre, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No